CLINICAL TRIAL: NCT01387789
Title: An Observational Study of Rheumatoid Arthritis Patients on Adalimumab to Evaluate Quality of Life Variables, Effects on Work Productivity and Functional Outcomes in Malaysia
Brief Title: A Study of Rheumatoid Arthritis Patients on Adalimumab to Evaluate Quality of Life Variables, Effects on Work Productivity and Functional Outcomes in Malaysia
Acronym: RELIVE
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-265
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Product Surveillance; Postmarketing
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Scheduled to start adalimumab therapy: Patients diagnosed with rheumatoid arthritis for at least 3 months that previously had not received prior anti-TNF agents.

SUMMARY:
An observational, non-interventional study on social, economic and quality-of-life outcomes of Adalimumab use in participants with moderate to severe active Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This study was designed to evaluate adalimumab therapy in Malaysia on participants' Quality of Life (QoL) using non-invasive epidemiological methods like the Health Assessment Questionnaire - Disability Index (HAQ-DI), the Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS), and the Health Assessment Questionnaire Short Form 36 (SF-36). The primary objective of the study was to evaluate the changes in QoL outcomes in anti -TNF naïve Malaysian RA patients after 6 months of adalimumab treatment. The secondary objectives of this study were to evaluate the changes on QoL outcomes after 1 month and 3 months of adalimumab treatment; and provide an assessment of the safety and tolerability of adalimumab in anti TNF naïve Malaysian Rheumatoid Arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older with a diagnosis of Rheumatoid Arthritis for at least 3 months according to the American College of Rheumatology (ACR) criteria
* Patients who have not been instituted on any anti -Tumour Necrosis Factor (anti-TNF) agents prior to inclusion into this study (anti-TNF naïve patients). Only anti-TNF Naive Rheumatoid Arthritis patients who are scheduled to begin HUMIRA treatment, according to the relevant Summary of Product Characteristics, on the basis of their own physician's judgment (and on the current clinical practice), will be selected for inclusion in this study
* Patients not included in other clinical/observational trials
* Patients providing a written informed consent before the enrollment in the study

Exclusion Criteria:

* Refusal to participate in the study or to sign the informed consent
* Contraindications to adalimumab according to the terms of the local marketing authorization (label)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mogana Sivalingam, MD, Study Director — AbbVie
Locations (13):
- Malaysia (13):
  - Site Reference ID/Investigator# 36098, Batu Caves
  - Site Reference ID/Investigator# 57913, George Town
  - Site Reference ID/Investigator# 57914, Ipoh
  - Site Reference ID/Investigator# 57923, Johor Bahru
  - Site Reference ID/Investigator# 67602, Klang
  - Site Reference ID/Investigator# 57925, Kota Kinabalu
  - Site Reference ID/Investigator# 57916, Kuala Lumpur
  - Site Reference ID/Investigator# 57928, Kuantan
  - Site Reference ID/Investigator# 57924, Kuching
  - Site Reference ID/Investigator# 57927, Malacca
  - Site Reference ID/Investigator# 57915, Putrajaya
  - Site Reference ID/Investigator# 57926, Serdang
  - Site Reference ID/Investigator# 57922, Seremban

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scheduled to Start Adalimumab Therapy
Started | 71
Completed | 63
Not Completed | 8
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
Age, Customized [Number; unit: participants]
  <30 years of age | 4
  30-39 years of age | 18
  40-49 years of age | 16
  50-59 years of age | 26
  60-69 years of age | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 9
Region of Enrollment [Number; unit: participants]
  Malaysia | 71

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Health Assessment Questionnaire Disability Index (HAQ-DI) Scores From Baseline to 6 Months
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥ 0.22. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5. Negative mean changes from baseline in the overall score indicate improvement. Assessments were conducted at baseline and 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
units on a scale | -0.41 (0.79)

2. Primary Outcome: Change in Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS) Scores From Baseline to 6 Months
Description: The Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS) is a patient-reported questionnaire designed to assess the presence or absence of arthritis-related pain and its severity. It consists of a doubly anchored, horizontal VAS, that is scored from 0 (no pain) to 100 (severe pain). Decreases from baseline indicate improvement. Assessments were conducted at baseline and 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
centimeters | -0.49 (0.79)

3. Primary Outcome: Change in Health Assessment Questionnaire Short Form 36 (SF-36) Scores From Baseline to 6 Months
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). The standard recall period is four weeks. Increases from baseline indicate improvement. Assessments were conducted at baseline and 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
units on a scale
  Physical Component Summary | 16.06 (23.02)
  Mental Component Summary | 12.30 (18.21)

4. Secondary Outcome: Change in Overall Health Assessment Questionnaire Disability Index (HAQ-DI) Scores From Baseline to 1 Month
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥0.22. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5. Negative mean changes from baseline in the overall score indicate improvement. Assessments were conducted at baseline and 1 month.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
units on a scale | -0.30 (0.52)

5. Secondary Outcome: Change in Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS) Scores From Baseline to 1 Month
Description: The Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS) is a patient-reported questionnaire designed to assess the presence or absence of arthritis-related pain and its severity. It consists of a doubly anchored, horizontal VAS, that is scored from 0 (no pain) to 100 (severe pain). Decreases from baseline indicate improvement. Assessments were conducted at baseline and 1 month.
Time Frame: Baseline and 1 month
Population: Participants with available data at this time point
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 70
centimeters | -0.46 (0.51)

6. Secondary Outcome: Change in Mean Health Assessment Questionnaire Short Form 36 (SF-36) Scores From Baseline to 1 Month
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). The standard recall period is four weeks. Increases from baseline indicate improvement. Assessments were conducted at baseline and 1 month.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
units on a scale
  Physical Component Summary | 11.46 (16.50)
  Mental Component Summary | 6.42 (13.56)

7. Secondary Outcome: Change in Overall Health Assessment Questionnaire Disability Index (HAQ-DI) Scores From Baseline to 3 Months
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥0.22. HAQ remission indicating normal physical function is defined by HAQ-DI < 0.5. Negative mean changes from baseline in the overall score indicate improvement. Assessments were conducted at baseline and 3 months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
units on a scale | -0.38 (0.69)

8. Secondary Outcome: Change in Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS) Scores From Baseline to 3 Months
Description: The Health Assessment Questionnaire Visual Analog Scale (HAQ-VAS) is a patient-reported questionnaire designed to assess the presence or absence of arthritis-related pain and its severity. It consists of a doubly anchored, horizontal VAS, that is scored from 0 (no pain) to 100 (severe pain). Decreases from baseline indicate improvement. Assessments were conducted at baseline and 3 months.
Time Frame: Baseline and 3 months
Population: Participants with available data at this time point
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 70
centimeters | -0.48 (0.72)

9. Secondary Outcome: Change in Health Assessment Questionnaire Short Form 36 (SF-36) Scores From Baseline to 3 Months
Description: The Health Assessment Questionnaire Short Form 36 (SF-36) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Items 5-8 primarily contribute to the mental component summary score (MCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best"). The standard recall period is four weeks. Increases from baseline indicate improvement. Assessments were conducted at baseline and 3 months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Scheduled to Start Adalimumab Therapy
Number analyzed (Participants) | 71
units on a scale
  Physical Component Summary | 14.19 (20.54)
  Mental Component Summary | 8.77 (15.55)

ADVERSE EVENTS:
Time Frame: SAEs were collected from the time the physician obtained the patient's informed consent until 30 days or 5 half-lives following the last dose of physician-prescribed treatment, an average of 250 days.
Arm/Group | Scheduled to Start Adalimumab Therapy
Serious Adverse Events (participants affected / at risk) | 13/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Scheduled to Start Adalimumab Therapy (N=71)
Anemia (Blood and lymphatic system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Pyrexia (General disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1
Antibiotic prophylaxis (Surgical and medical procedures) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.